CLINICAL TRIAL: NCT06264544
Title: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial to Evaluate the Efficacy of a Zinc, Selenium, and L-Tyrosine Supplement in the Prevention of Thyrotoxicosis in Subjects With r25191G/A SEPP1 Polymorphism
Brief Title: Trial to Evaluate the Efficacy of a Zinc, Selenium, and L-Tyrosine Supplement in the Prevention of Thyrotoxicosis in Subjects With r25191G/A SEPP1 Polymorphism
Acronym: ZEST-PREP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: S.LAB (SOLOWAYS) (Other)
Collaborators: Center of New Medical Technologies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SW006
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Thyrotoxicosis
Keywords: Thyrotoxicosis Prevention; SEPP1 Polymorphism; Zinc, Selenium, and L-Tyrosine Supplementation; supplementation; Nutrigenomics; Thyroid Peroxidase Antibodies (TPOAb)
MeSH Terms: conditions — Thyrotoxicosis | interventions — Zinc; Selenium; Tyrosine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- zinc, selenium, and L-tyrosine supplementation (Experimental)
  Interventions: Dietary Supplement: zinc, selenium, and L-tyrosine in SEPP1
- placebo group (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: zinc, selenium, and L-tyrosine in SEPP1 — zinc, selenium, and L-tyrosine in SEPP1 polymorphism
  Arms: zinc, selenium, and L-tyrosine supplementation
Other: Placebo — placebo comparator in SEPP1 polymorphism group
  Arms: placebo group

SUMMARY:
This randomized, double-blind, placebo-controlled trial evaluates the efficacy of a zinc, selenium, and L-tyrosine supplement in preventing thyrotoxicosis among adults aged 18-85 with elevated TPOAb levels and the r25191G/A SEPP1 polymorphism. The study excludes those with thyroid disease, pregnant/breastfeeding women, and individuals allergic to the supplement. Key endpoints include changes in thyroid antibodies and hormones over a 6-month period. With an estimated sample size of 150 participants per group, accounting for a 20% dropout rate, the trial seeks to demonstrate the supplement's potential in reducing thyrotoxicosis risk through a genetically-informed approach.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed presence of one or more specified gene polymorphism r25191G/A SEPP1
* TPOAb levels > 300 IU/mL

Exclusion Criteria:

* Age < 18 years and >85
* Pregnant or breastfeeding woman
* Subjects with allergy to any of the supplementation component patients with any established diagnosis of thyroid disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Percent change of Thyroid Peroxidase Antibodies (TPOAb) in subjects with r25191 SEPP1 polymorphism | 6 months

SECONDARY OUTCOMES:
Percent change in Thyroglobulin Antibodies (TgAb) in subjects with r25191 SEPP1 polymorphism | 6 months
Free Thyroxine (Free T4) change in subjects with r25191 SEPP1 polymorphism | 6 months
Free Triiodothyronine (Free T3) change in subjects with r25191 SEPP1 polymorphism | 6 months
Thyroid Receptor Antibodies (TRAb) change in subjects with r25191 SEPP1 polymorphism | 6 months
TSH Receptor Antibodies (TSHR-Ab) change in subjects with r25191 SEPP1 polymorphism | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Center of New Medical Technologies, Novosibirsk, Novosibisk Region, Russia

IPD SHARING:
Plan to Share IPD: No